CLINICAL TRIAL: NCT05318300
Title: Assessment of the Effect of Cow's Milk Protein-based Formulas for Infants in the Management of Moderate to Severe aTOPic Dermatitis in Infants Aged Less Than 18 Months
Brief Title: Evaluation of an Adapted Formula on Atopic Dermatitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP2018-EFITOP
Record Dates: First submitted 2022-03-18; First posted 2022-04-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tested formula LP-2018 (Experimental): infant formula containing fibers
  Interventions: Dietary Supplement: tested formula with fiber
- Placebo formula CT-2018 (Placebo Comparator): infant formula without fibers
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: tested formula with fiber — formula containing fibers
  Arms: Tested formula LP-2018
Dietary Supplement: Control — formula without fiber
  Arms: Placebo formula CT-2018

SUMMARY:
The aim of this study is to show the efficiency of a new infant formula containing fiber on the management of moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
The study is double blind randomized where the new formula is compared to a placebo during 3 months followed by a period of 3 months optional. During this period of time, all infant include in the study will be fed with the study formula.

ELIGIBILITY:
Inclusion Criteria:

* Aged below 18 month
* Having an atopic dermatitis diagnosed according to the United Kingdom Working Party - Having an Eczema Area Severity Index (EASI) between 7.1 and 50.0
* Whose parents gave their informed consent

Exclusion Criteria:

* systemic corticotherapy
* antihistamine
* use of dermocorticoide and/or antibiotics within 15 days
* symptoms of cutaneous infection
* Past anaphylactic shock
* cow's milk, soya or fish allergy
* Exclusive or predominant breast feediing (more than one feeding/day)
* Consumption of less than 500 ml per day
* Participation to another trial.

Ages: 1 Month to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2022-05-24 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
EASI (Eczema Area Severity Index) score after 90 days. | 90 days
  evolution of the EASI score between day 0 to day 90. The score range is between 0 (no eczema) and 72 (highest score of eczema)

SECONDARY OUTCOMES:
EASI (Eczema Area Severity Index) score after 30 days. | 30 days
  evolution of the EASI score between day 0 to day 30. The score range is between 0 (no eczema) and 72 (highest score of eczema)
EASI (Eczema Area Severity Index) score after 60 days. | 60 days
  evolution of the EASI score between day 0 to day 60. The score range is between 0 (no eczema) and 72 (highest score of eczema)
EASI (Eczema Area Severity Index) score after 180 days. | 180 days
  evolution of the EASI score between day 0 to day 180. The score range is between 0 (no eczema) and 72 (highest score of eczema)
PO SCORAD (Patient Oriented-SCORing Atopic Dermatitis ) evolution | 30 days
  Area under the curve of PO SCORAD
PO SCORAD (Patient Oriented-SCORing Atopic Dermatitis ) evolution | 60 days
  Area under the curve of PO SCORAD
PO SCORAD (Patient Oriented-SCORing Atopic Dermatitis ) evolution | 90 days
  Area under the curve of PO SCORAD
PO SCORAD (Patient Oriented-SCORing Atopic Dermatitis ) evolution | 180 days
  Area under the curve of PO SCORAD
Skin dryness | 30 days
  Evolution of skin dryness evaluated by the investigator using the dryness scale of the PO SCORAD
Skin dryness | 60 days
  Evolution of skin dryness evaluated by the investigator using the dryness scale of the PO SCORAD
Skin dryness | 90 days
  Evolution of skin dryness evaluated by the investigator using the dryness scale of the PO SCORAD
Skin dryness | 180 days
  Evolution of skin dryness evaluated by the investigator using the dryness scale of the PO SCORAD
Itching | 30 days
  Evolution of itching evaluated by the investigator using an analogic visual scale
Itching | 60 days
  Evolution of itching evaluated by the investigator using an analogic visual scale
Itching | 90 days
  Evolution of itching evaluated by the investigator using an analogic visual scale
Itching | 180 days
  Evolution of itching evaluated by the investigator using an analogic visual scale
Quality of sleep (assessed by VAS) | 30 days
  Evalution of the quality of sleep by the investigator using an analogic visual scale (from 0 to 10) (0 means no sleeping troubles and 10 mens very important troubles)
Quality of sleep (assessed by VAS) | 60 days
  Evalution of the quality of sleep by the investigator using an analogic visual scale (from 0 to 10) (0 means no sleeping troubles and 10 mens very important troubles)
Quality of sleep (assessed by VAS) | 90 days
  Evalution of the quality of sleep by the investigator using an analogic visual scale (from 0 to 10) (0 means no sleeping troubles and 10 mens very important troubles)
Quality of sleep (assessed by VAS) | 180 days
  Evalution of the quality of sleep by the investigator using an analogic visual scale (from 0 to 10) (0 means no sleeping troubles and 10 mens very important troubles)
Sleep time | 30 days
  Evaluation of the duration of sleep by parents
Sleep time | 60 days
  Evaluation of the duration of sleep by parents
Sleep time | 90 days
  Evaluation of the duration of sleep by parents
Sleep time | 180 days
  Evaluation of the duration of sleep by parents
IDQoL (Infant's Dermatitis Quality of Life) | 90 days
  Evaluation of the infant's quality of life through the IDQoL (Infant's Dermatitis Quality of Life)
Use of topical dermocorticoids | 30 days
  The quantity and class of dermocorticoids used will be evaluated
Use of topical dermocorticoids | 60 days
  The quantity and class of dermocorticoids used will be evaluated
Use of topical dermocorticoids | 90 days
  The quantity and class of dermocorticoids used will be evaluated
Use of topical dermocorticoids | 180 days
  The quantity and class of dermocorticoids used will be evaluated
Atopic dermatitis flare | 30 days
  The number of flare will be evaluated
Atopic dermatitis flare | 60 days
  The number of flare will be evaluated
Atopic dermatitis flare | 90 days
  The number of flare will be evaluated
Atopic dermatitis flare | 180 days
  The number of flare will be evaluated
Weight | 30 days
  Weight evolution
Weight | 60 days
  Weight evolution
Weight | 90 days
  Weight evolution
Weight | 180 days
  Weight evolution
Length/Height | 30 days
  Length/Height evolution
Length/Height | 60 days
  Length/Height evolution
Length/Height | 90 days
  Length/Height evolution
Length/Height | 180 days
  Length/Height evolution
Regurgitations | Day 30
  Evolution of the daily number of regurgitations
Regurgitations | Day 60
  Evolution of the daily number of regurgitations
Regurgitations | Day 90
  Evolution of the daily number of regurgitations
Regurgitations | Day 180
  Evolution of the daily number of regurgitations
Stool's frequency | Day 30
  Evolution of the number of stools per day through a qualitative scale
Stool's frequency | Day 60
  Evolution of the number of stools per day through a qualitative scale
Stool's frequency | Day 90
  Evolution of the number of stools per day through a qualitative scale
Stool's frequency | Day 180
  Evolution of the number of stools per day through a qualitative scale
Stool's consistency | Day 30
  Evolution of the stool's consistency using the Brussels Infant and Toddler Stool Scale
Stool's consistency | Day 60
  Evolution of the stool's consistency using the Brussels Infant and Toddler Stool Scale
Stool's consistency | Day 90
  Evolution of the stool's consistency using the Brussels Infant and Toddler Stool Scale
Stool's consistency | Day 180
  Evolution of the stool's consistency using the Brussels Infant and Toddler Stool Scale
Gas, bloating | Day 30
  Evolution of presence/absence of gas, bloating
Gas, bloating | Day 60
  Evolution of presence/absence of gas, bloating
Gas, bloating | Day 90
  Evolution of presence/absence of gas, bloating
Gas, bloating | Day 180
  Evolution of presence/absence of gas, bloating
Satisfaction of the parents | Day 30
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the parents | Day 60
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the parents | Day 90
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the parents | Day 180
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the investigator | Day 30
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the investigator | Day 60
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the investigator | Day 90
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas
Satisfaction of the investigator | Day 180
  Different levels of satisfaction (from bad to good/very good) on the use and efficiency of study formulas

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne Cahn-Sellem, Principal Investigator — Private Practice; Sebastien Barbarot, Study Chair — Hotel Dieu Hospital, Nantes, France; Elena Bradatan, Principal Investigator — Private Practice
Locations (3):
- Belgium (2):
  - Center_13, Namur
  - Center_14, Thuin
- Center_05, Nice, France

IPD SHARING:
Plan to Share IPD: No